CLINICAL TRIAL: NCT06917612
Title: Normal Diagnostic Laparoscopy Versus Negative Appendectomy in Patients With a Normal Appendix Undergoing Laparoscopic Surgery for Suspected Appendicitis: a Target Trial
Brief Title: Preserving or Resecting the Normal Appendix in Patients Undergoing Laparoscopy Surgery for Suspected Appendicitis
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: Danish Institute for Public Health (Other)
Responsible Party: Principal Investigator, Siv Fonnes, Researcher, MD, PhD, Herlev Hospital
Other Study IDs: HEH-SF-03
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Acute Appendicitis; Abdominal Pain (AP); Diagnostic Laparoscopy; Laparoscopic Appendectomy; Neoplasms
MeSH Terms: conditions — Appendicitis; Abdominal Pain; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal diagnostic laparoscopy group: The appendix is left in situ, e.g. not resected and no other surgical procedure is needed to treat other diseases, identified through both the nationwide Danish National Patient Register and Danish Pathology Data Bank
  Interventions: Procedure: Normal diagnostic laparoscopy
- Negative appendectomy group: The appendix is resected but is without histopathological inflammation and no other surgical resection is needed to treat other diseases, identified through both the nationwide Danish National Patient Register and Danish Pathology Data Bank
  Interventions: Procedure: Negative appendectomy

INTERVENTIONS:
Procedure: Normal diagnostic laparoscopy — The appendix is left in situ e.g., not resected and no other surgical resection is needed to treat other diseases
  Groups: Normal diagnostic laparoscopy group
Procedure: Negative appendectomy — The appendix is resected but is without histopathological-confirmed inflammation and no other surgical resection is needed to treat other diseases
  Groups: Negative appendectomy group

SUMMARY:
When appendicitis is suspected, patients are typically planned for emergency surgery preferably using a laparoscopic approach. Up to 20% of these patients will have a normal appendix, thus not suffering from appendicitis. Surgeons can either perform a normal diagnostic laparoscopy (leave the appendix in situ) or perform a negative appendectomy (resect the normal appendix). International guidelines recommend negative appendectomy based on weak evidence due to the risk of appendix cancer, but some countries and researchers advocate against negative appendectomy as these patients may experience more harm than if the appendix is left in situ. There are limited national guidelines and the decision is often left to the operating surgeon. Surgeons performing negative appendectomies argue that these prevent microappendicitis and the risk of a subsequent episode of appendicitis. As appendix cancers are rare, and a randomised controlled trial including this subgroup of patients with normal appendices undergoing emergency surgery for suspected appendicitis is unfeasible, an emulated target trial is planned.

This target trial aims to evaluate the effect of a normal diagnostic laparoscopy versus negative appendectomy during laparoscopic surgery for suspected appendicitis regarding cancer in the appendix and other complications such as death, reoperation, and readmission.

DETAILED DESCRIPTION:
The target trial emmulates an unfeasible randomised controlled trial by using observational data to investigate the two treatment strategies (two groups) normal diagnostic laparoscopy versus negative appendectomy when a normal appendix is seen during surgery for suspected appendicitis. The assignment to the treatment strategies during surgery for suspected appendicitis is treated as randomised within the levels of the following baseline covariates; sex, age, year of index surgery, and hospital through inverse probability weighting. We will analyse data according to treatment assignment at baseline (intention-to-treat). Because the treatment strategies in this target trial are surgical, all participants will adhere to the surgical treatment strategy: neither a normal diagnostic laparoscopy nor a negative appendectomy at index surgery can be reversed. However, both may be followed by a reoperation, e.g., a new normal diagnostic laparoscopy or a laparoscopic appendectomy (for suspected appendicitis or stump appendicitis). However, this will not influence analyses but be recorded as an outcome.

As inverse probability weighting has been applied, no further adjustment in the pre-specified analyses below is needed.

The continuous outcome, delay of cancer diagnosis for the normal diagnostic laparoscopy group, will be descriptively reported as mean (SD) or median (IQR).

For dichotomous outcomes, the following analyses are planned:

* Kaplan-Meier curves for each group
* Incidence proportion (risk) including 95% CI for each group
* Relative risk
* Risk difference
* Number needed to treat
* Number needed to harm
* Test chi-square

ELIGIBILITY:
Inclusion Criteria:

* All ages and sexes
* Undergoing laparoscopic surgery for suspected appendicitis from 2005 to 2021
* Resected appendix without inflammation e.g., without appendicitis

Exclusion Criteria:

* Previous resection of the appendix (e.g., previous appendectomy, or resection of the gut including the appendix before January 1, 2005) based on data from surgical codes in the Danish National Patient Register
* Unable to be tracked in the Danish registers, such as a replacement personal identification number, or for those not residing in Denmark based on data from the Civil Registration System
* Diagnostic codes indicating appendix cancer at index surgery (C181), thus, not operated for suspected appendicitis
* Laparoscopic appendectomy converted to open surgery or other surgical procedures conducted contaminated with laparoscopic appendectomy, indicated a need for other surgical interventions because of disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages undergoing laparoscopic surgery for suspected appendicitis, as recorded in the nationwide Danish National Patient Register, are identified via diagnostic and surgical codes. Information on negative appendectomies is retrieved from the nationwide register of the Danish Pathology Data Bank.
  We will use inverse probability weighting to adjust for and minimise bias derived from an imbalance in baseline covariates (sex, age, year of surgery, and hospital).
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Cancer in the appendix | 2 years
  Histopathologically verified cancer in the appendix (primary or metastasis) in the nationwide register the Danish Pathology Data Bank e.g., SNOMED morphology codes for cancer (M8**** or M9****) in relation to the topography code of the appendix (T66000)
Appendix cancer | 2 years
  Histopathologically verified appendix cancer (primary) in the nationwide register the Danish Pathology Data Bank e.g., SNOMED morphology codes for cancer (M8**** or M9****) in relation to the topography code of the appendix (T66000)

SECONDARY OUTCOMES:
Delay in diagnosis of cancer | 2 years
  Time from index normal diagnostic laparoscopy to histopathologically verified cancer in the appendix in the nationwide register Danish Pathology Data Bank, e.g., SNOMED morphology codes for cancer (M8**** or M9****) in relation to the topography code of the appendix (T66000)
Death | 2 years
  All-cause death registered in the nationwide The Civil Registration System
Any reoperation | 1 year
  Any reoperations registered in the nationwide Danish National Patient Register
Abdominal reoperation | 1 year
  Abdominal reoperations registered in the nationwide Danish National Patient Register e.g., with surgical codes KJ*** (gastrointestinal tract), KK*** (urological), or KL***(gynecological)
Resected appendix | 2 years
  Histopathological record of an appendix in the nationwide register the Danish Pathology Data Bank e.g., record with topography code of the appendix (T66000) after index surgery, including subdivision of morphology codes into appendicitis, negative appendectomy, appendix cancer, and other
Readmission | 1 year
  Any readmissions registered in the nationwide Danish National Patient Register, including subdivisions into diagnostic codes relating to different diseases

OTHER OUTCOMES:
Subgroup analysis for outcomes at 1 year follow-up | 1 year
  Subgroup analyses of all primary and secondary outcomes at the time-point 1 year after index surgery, including 100% of the included participants in the target trial
Subgroup analysis for outcomes at 2 years follow-up | 2 year
  Subgroup analyses of all primary and secondary outcomes at the time-point 2 years after index surgery, including 75% to <100% of the included participants in the target trial
Subgroup analysis for outcomes at 5 years follow-up | 5 year
  Subgroup analyses of all primary and secondary outcomes at the time-point 5 years after index surgery, including as few as 75% of the included participants in the target trial
Sensitivity analysis on comorbidity | 1 year
  For the secondary outcomes (death (2 years), reoperation, and readmission), confounding due to comorbidity will be explored for patients undergoing index surgery from January 1, 2010, and onwards, thus, allowing for calculating Charlson Comorbidity Index based data in the nationwide Danish National Patient Register from 5 years before to index surgery
Sensitivity analysis on umeasured confounding | 2 years
  For the primary outcomes, unmeasured confounding e.g., due to preoperative imaging or perioperative macroscopic suspicion of cancer, will be addressed by calculating the E value

CONTACTS AND LOCATIONS:
Overall Officials: Siv Fonnes, MD, PhD, Principal Investigator — Herlev Hospital

IPD SHARING:
Plan to Share IPD: No
The researchers have access to pseudonymised data provided by Statistics Denmark, and according to their rules and guidelines on transfer and data security (https://www.dst.dk/en/TilSalg/data-til-forskning/regler-og-datasikkerhed/regler-for-hjemtagelse-af-analyseresultater) information on individual level cannot be transferred outside Statistics Denmark's researcher machines.